CLINICAL TRIAL: NCT05441436
Title: Identification of Needs and Neuropsychological and Biopsychosocial Evolution in the Pre/Post-transplant and 6-month Follow-up Phases in Pediatric Population (the TransplantKIDS Mental Health Project)
Brief Title: Neuropsychological and Biopsychosocial Evolution During Pediatric Transplantation: Pre/Post-stages and at 6 Months
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Universitario La Paz (Other)
Collaborators: University of Malaga (Other)
Responsible Party: Principal Investigator, Dr. Eduardo Fernández-Jiménez, Principal Investigator, Hospital Universitario La Paz
Other Study IDs: 5223
Record Dates: First submitted 2022-06-13; First posted 2022-07-01 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Transplant-Related Disorder
Keywords: Pediatric Solid Organ Transplant; Pediatric Allogeneic Hematopoietic Transplant; Neuropsychology; Biopsychosocial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Allogeneic hematopoietic stem cell transplantation: Patients in waiting list for and after allogeneic hematopoietic stem cell transplantation.
  Interventions: Procedure: Allogeneic hematopoietic stem cell transplantation
- Solid organ transplantation: Patients in waiting list for and after solid organ transplantation.
  Interventions: Procedure: Solid organ transplantation

INTERVENTIONS:
Procedure: Allogeneic hematopoietic stem cell transplantation — Allogeneic hematopoietic stem cell transplantation
  Groups: Allogeneic hematopoietic stem cell transplantation
Procedure: Solid organ transplantation — Solid organ transplantation
  Groups: Solid organ transplantation

SUMMARY:
This pioneering prospective observational study aims to examine biopsychosocial and neuropsychological functioning, care needs and predictors of therapeutic adherence in children/adolescents in pre/post-surgical transplant (solid organ or allogeneic haematopoietic stem cell) phases. Hypothesis: H1. Differences in biopsychosocial and neuropsychological functioning and adherence will be observed between transplant types; H2. Executive functioning will mediate the relationship between anxiety, sleep disturbance and pain intensity/interference and adherence; H3. There will be a significant improvement in different neuropsychological indicators 6 months post-transplantation. Sample: patients (8-18 years) extracted by non-probabilistic sampling, estimating a sample size of 60 patients (30 for each type of transplant, organ and haematopoietic) from Hospital Universitario La Paz (Madrid). Individual pre/post-surgical assessments will be carried out (after 2 and 4 weeks), as well as at 6 months post-transplant, both in person (neurocognitive) and through the secure platform REDCap (completed by patients and their legal guardians). Finally, focus groups will be conducted among patients, their relatives and medical-surgical professionals to identify barriers to therapeutic adherence and unmet care needs during the pre-, peri- and post-surgical process.

ELIGIBILITY:
Inclusion Criteria:

* Spanish as mother tongue or a very high level of Spanish in order to understand their participation in the study, as well as to be able to complete the measurement instruments.

Exclusion Criteria:

* Diagnosis of intellectual disability, autism spectrum disorder or acquired brain damage.
* Diagnosis of uncontrolled/stabilised comorbid disease, independent of the disease motivating the transplantation process.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Potential participants will be all children and adolescents in the imminent phase of being included in the waiting list for a transplant of any solid organ (single or combined), or allogeneic haematopoietic stem cell.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-05-26 (Actual); Primary Completion 2025-05-26 (Estimated); Study Completion 2025-05-26 (Estimated)

PRIMARY OUTCOMES:
Initial survey created ad hoc | Baseline
  Both sociodemographic variables (sex, age, patient's level of studies, parents' level of studies) and clinical variables (current pharmacological treatment - active ingredient and dose) will be collected.
Behavior Rating Inventory of Executive Function - 2 (BRIEF-2) | Baseline
  A 63-item questionnaire that assesses patient's executive functions (completed by parents). Higher scores in each domain indicate a worse outcome. Spanish norms in T scores (Mean = 50; standard deviation = 10).
Behavior Rating Inventory of Executive Function - 2 (BRIEF-2) | 6 months
  A 63-item questionnaire that assesses patient's executive functions (completed by parents). Higher scores in each domain indicate a worse outcome. Spanish norms in T scores (Mean = 50; standard deviation = 10).
Spanish version of the California Verbal Learning Test for children (TAVECI) | Baseline
  Assessment of verbal memory in children 3 to 16 years old by the maximum number of remembered elements.
Spanish version of the California Verbal Learning Test (TAVEC) | Baseline
  Assessment of verbal memory for adolescents 16 to 18 years old by the maximum number of remembered elements.
Spanish version of the California Verbal Learning Test for children (TAVECI) | 6 months
  Assessment of verbal memory in children 3 to 16 years old by the maximum number of remembered elements.
Spanish version of the California Verbal Learning Test (TAVEC) | 6 months
  Assessment of verbal memory for adolescents 16 to 18 years old by the maximum number of remembered elements.
Conners Continuous Auditory Test of Attention (CATA) | Baseline
  It measures auditory sustained attention. Omissions and commissions are measured for 5 different dimensions: inattentiveness, impulsivity, sustained attention, auditory laterality and auditory mobility.
Conners Continuous Auditory Test of Attention (CATA) | 4 weeks
  It measures auditory sustained attention. Omissions and commissions are measured for 5 different dimensions: inattentiveness, impulsivity, sustained attention, auditory laterality and auditory mobility.
Conners Continuous Auditory Test of Attention (CATA) | 6 months
  It measures auditory sustained attention. Omissions and commissions are measured for 5 different dimensions: inattentiveness, impulsivity, sustained attention, auditory laterality and auditory mobility.
Test of Nonverbal Intelligence, Fourth Edition (TONI-4) form A | Baseline
  It assesses intellectual functioning free of cultural influences by the total number of items achieved.
Test of Nonverbal Intelligence, Fourth Edition (TONI-4) form B | 6 months
  It assesses intellectual functioning free of cultural influences by the total number of items achieved.
Digit span subtests from the Wechsler Intelligence Scale for Children, Fifth Edition (WISC-V) or the Wechsler Adult Intelligence Scale, Fourth Edition (WAIS-IV): Forward, Backward and Sequencing subtests | Baseline
  It evaluates span of immediate recall and verbal working memory by the total number of items achieved and the maximum number of remembered elements.
Digit span subtests from the Wechsler Intelligence Scale for Children, Fifth Edition (WISC-V) or the Wechsler Adult Intelligence Scale, Fourth Edition (WAIS-IV): Forward, Backward and Sequencing subtests | 4 weeks
  It evaluates span of immediate recall and verbal working memory by the total number of items achieved and the maximum number of remembered elements.
Digit span subtests from the Wechsler Intelligence Scale for Children, Fifth Edition (WISC-V) or the Wechsler Adult Intelligence Scale, Fourth Edition (WAIS-IV): Forward, Backward and Sequencing subtests | 6 months
  It evaluates span of immediate recall and verbal working memory by the total number of items achieved and the maximum number of remembered elements.
Vocabulary subtest from the Wechsler Intelligence Scale for Children, Fifth Edition (WISC-V) or the Wechsler Adult Intelligence Scale, Fourth Edition (WAIS-IV) | Baseline
  It measures semantic memory by the total number of items achieved.
Vocabulary subtest from the Wechsler Intelligence Scale for Children, Fifth Edition (WISC-V) or the Wechsler Adult Intelligence Scale, Fourth Edition (WAIS-IV) | 6 months
  It measures semantic memory by the total number of items achieved.
Symbol Digit Modalities Test (SDMT) | Baseline
  It assesses processing speed by the total number of items achieved.
Symbol Digit Modalities Test (SDMT) | 4 weeks
  It assesses processing speed by the total number of items achieved.
Symbol Digit Modalities Test (SDMT) | 6 months
  It assesses processing speed by the total number of items achieved.
The Rey-Osterrieth Complex Figure (ROCF) test | Baseline
  It measures viso-constructive organisational ability and immediate and delayed visual recall. One point is awarded for each component that is properly reproduced.
The Rey-Osterrieth Complex Figure (ROCF) test | 6 months
  It measures viso-constructive organisational ability and immediate and delayed visual recall. One point is awarded for each component that is properly reproduced.
Fluency Verbal Test (TFV) | Baseline
  It assesses linguistic-executive functions such as phonological fluency and semantic fluency. One point is awarded for each word that is correctly produced.
Fluency Verbal Test (TFV) | 6 months
  It assesses linguistic-executive functions such as phonological fluency and semantic fluency. One point is awarded for each word that is correctly produced.
Behavioral Assessment System for Children - 3 (BASC-3) | Baseline
  It measures patients' emotional and behavioural problems, both in its version by the patient's legal guardians and self-reported by the patient. It is an 139-item report, rated on a 4-point frequency Likert scale. High scores indicate problematic levels of functioning. Spanish norms in T scores (Mean = 50; standard deviation = 10).
Behavioral Assessment System for Children - 3 (BASC-3) | 6 months
  It measures patients' emotional and behavioural problems, both in its version by the patient's legal guardians and self-reported by the patient. It is an 139-item report, rated on a 4-point frequency Likert scale. High scores indicate problematic levels of functioning. Spanish norms in T scores (Mean = 50; standard deviation = 10).
Brief Pain Inventory (BPI) | Baseline
  This 10-item questionnaire includes questions (from 0 to 10 referring to the last 7 days) covering two dimensions: pain intensity (worst and mildest pain in the week, average pain, and current pain), and pain interference (with general activity, mood, walking, school, sleep, as well as enjoyment of life). Higher scores on a Likert scale from 0-10 indicate more pain.
Brief Pain Inventory (BPI) | 2 weeks
  This 10-item questionnaire includes questions (from 0 to 10 referring to the last 7 days) covering two dimensions: pain intensity (worst and mildest pain in the week, average pain, and current pain), and pain interference (with general activity, mood, walking, school, sleep, as well as enjoyment of life). Higher scores on a Likert scale from 0-10 indicate more pain.
Brief Pain Inventory (BPI) | 4 weeks
  This 10-item questionnaire includes questions (from 0 to 10 referring to the last 7 days) covering two dimensions: pain intensity (worst and mildest pain in the week, average pain, and current pain), and pain interference (with general activity, mood, walking, school, sleep, as well as enjoyment of life). Higher scores on a Likert scale from 0-10 indicate more pain.
Brief Pain Inventory (BPI) | 6 months
  This 10-item questionnaire includes questions (from 0 to 10 referring to the last 7 days) covering two dimensions: pain intensity (worst and mildest pain in the week, average pain, and current pain), and pain interference (with general activity, mood, walking, school, sleep, as well as enjoyment of life). Higher scores on a Likert scale from 0-10 indicate more pain.
Adolescent Insomnia Questionnaire (AIQ) | Baseline
  It is a 13-item questionnaire whose original version is in English. In the present study, this questionnaire will be adapted and validated into Spanish. Higher scores on a Likert scale from 0-4 indicate more insomnia.
Adolescent Insomnia Questionnaire (AIQ) | 2 weeks
  It is a 13-item questionnaire whose original version is in English. In the present study, this questionnaire will be adapted and validated into Spanish. Higher scores on a Likert scale from 0-4 indicate more insomnia.
Adolescent Insomnia Questionnaire (AIQ) | 4 weeks
  It is a 13-item questionnaire whose original version is in English. In the present study, this questionnaire will be adapted and validated into Spanish. Higher scores on a Likert scale from 0-4 indicate more insomnia.
Adolescent Insomnia Questionnaire (AIQ) | 6 months
  It is a 13-item questionnaire whose original version is in English. In the present study, this questionnaire will be adapted and validated into Spanish. Higher scores on a Likert scale from 0-4 indicate more insomnia.
Pediatric Sleep Disturbances Short Form (PROMIS) | Baseline
  A 4-item questionnaire that assesses problems with sleep reconciliation and sleep maintenance in the last 7 days. Higher scores on a Likert scale from 1-5 indicate worse sleep.
Pediatric Sleep Disturbances Short Form (PROMIS) | 2 weeks
  A 4-item questionnaire that assesses problems with sleep reconciliation and sleep maintenance in the last 7 days. Higher scores on a Likert scale from 1-5 indicate worse sleep.
Pediatric Sleep Disturbances Short Form (PROMIS) | 4 weeks
  A 4-item questionnaire that assesses problems with sleep reconciliation and sleep maintenance in the last 7 days. Higher scores on a Likert scale from 1-5 indicate worse sleep.
Pediatric Sleep Disturbances Short Form (PROMIS) | 6 months
  A 4-item questionnaire that assesses problems with sleep reconciliation and sleep maintenance in the last 7 days. Higher scores on a Likert scale from 1-5 indicate worse sleep.
Simplified Medication Adherence Questionnaire (SMAQ) | Baseline
  A 6-item self-report that measures adherence to medication. For items 1-4 yes or no answers are required. Item 5 requires a multiple choice answer in terms of frequency (5 different options are provided). Item 6 requires a number input. The final score is a dichotomous variable: non-adherent versus adherent patient.
Simplified Medication Adherence Questionnaire (SMAQ) | 2 weeks
  A 6-item self-report that measures adherence to medication. For items 1-4 yes or no answers are required. Item 5 requires a multiple choice answer in terms of frequency (5 different options are provided). Item 6 requires a number input. The final score is a dichotomous variable: non-adherent versus adherent patient.
Simplified Medication Adherence Questionnaire (SMAQ) | 4 weeks
  A 6-item self-report that measures adherence to medication. For items 1-4 yes or no answers are required. Item 5 requires a multiple choice answer in terms of frequency (5 different options are provided). Item 6 requires a number input. The final score is a dichotomous variable: non-adherent versus adherent patient.
Simplified Medication Adherence Questionnaire (SMAQ) | 6 months
  A 6-item self-report that measures adherence to medication. For items 1-4 yes or no answers are required. Item 5 requires a multiple choice answer in terms of frequency (5 different options are provided). Item 6 requires a number input. The final score is a dichotomous variable: non-adherent versus adherent patient.

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Fernández-Jiménez, PhD, Principal Investigator — Hospital Universitario La Paz
Locations (2):
- Spain (2):
  - Hospital Universitario La Paz. Hospital infantil, Madrid
  - University of Málaga, Málaga

REFERENCES:
- [Derived] Garrido-Bolton J, Alcami-Pertejo M, de la Vega R, Hernandez-Oliveros F, Perez-Martinez A, Bravo-Ortiz MF, Fernandez-Jimenez E. Neuropsychological and biopsychosocial evolution, therapeutic adherence and unmet care needs during paediatric transplantation: study protocol of a mixed-methods design (observational cohort study and focus groups) - the TransplantKIDS mental health project. Front Psychol. 2024 Feb 21;15:1308418. doi: 10.3389/fpsyg.2024.1308418. eCollection 2024. PMID 38449767